CLINICAL TRIAL: NCT02267941
Title: Food and Drug Administration in China
Brief Title: Risk Factors for Aortic Dissection in the Chinese Patients
Status: Completed | Type: Observational
Sponsor: General Hospital of Beijing PLA Military Region (Other)
Responsible Party: Principal Investigator, Yang Li, Doctor, General Hospital of Beijing PLA Military Region
Other Study IDs: GHBeijing-20140702
Record Dates: First submitted 2014-09-20; First posted 2014-10-20 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2013-12

CONDITIONS: Persistent Blood Flow in False Lumen of Aortic Dissection
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- case: Diagnosis of aortic dissection was based on history and physical examination, and confirmed by imaging, visualization at surgery, and/or postmortem examination. According to the Stanford classification system, type A aortic dissection was defined as any dissection that involves the ascending aorta and type B as any that does not. Acute stage was confined to initial 14 days after symptom onset. Simple aortic aneurysm and pseudoaneurysm were excluded. Surgical and endovascular treatments were the main interventions and performed in the case group.
  Interventions: Other: observation
- control: As the control group, 2760 patients without AD were obtained from the hospitalized patients in the same period. Types of disease in the control group included congenital heart disease (632), coronary heart disease (467), adult valve disease (375), pulmonary artery hypertension (292), appendicitis (234), pneumonia (197), fracture (189), intestinal polyps (167), gallstone (156), esophagus cancer (51). Patients in the control group were derived from Department of Cardiovascular Surgery, Department of General Surgery, Department of Thoracic Surgery, and Department of Respiration, respectively.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — Data were collected by a disigned form. Statistic software was used to analyze clinical data.

SUMMARY:
To evaluate epidemiological features of risk factors for aortic dissection (AD) in Chinese patients.

DETAILED DESCRIPTION:
Aortic dissection (AD) is a life-threatening cardiovascular disease with high mortality. Without optimal treatment, approximately 50% of patients die within one week of the onset of symptoms, and 80% die within 2 weeks. With the change of life-style and the development of diagnostic technology, the incidence and detection rate of AD were increasing in China recently. However, the cause remains unclear. Studies showed that AD were associated with some risk factors, such as hypertension, connective tissue disease, iatrogenic injury, drug, pregnancy, etc. It is reported that two thirds patients with AD had a history of hypertension; 50% patients aged <40 years were accompanied with hereditary Marfan syndrome; 13～19% had a familial history of aortic aneurysm or dissection. These epidemiological data were obtained from Caucasian population, however, such information was not available for the Chinese population. Moreover, epidemiological investigation was absent in China, and the assessment of risk factors for AD was mainly referred to the studies from developed countries. Therefore, the aim of our study was to evaluate epidemiological features of risk factors for AD in Chinese patients using 3045 individuals from the 15 major centers in China. We anticipated that this analysis would provide helpful information preventing and controlling AD in China.

ELIGIBILITY:
Inclusion Criteria:

* Aortic dissection
* Acute stage

Exclusion Criteria:

-Simple aortic aneurysm and pseudoaneurysm were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January, 2011 and December, 2012, we collected 3045 patients with AAD (1668 with type A and 1377 with type B) from 15 major centers in China as the case group. As the control group, 2760 patients without AD were obtained from the hospitalized patients in the same period.
Sampling Method: Probability Sample
Enrollment: 3045 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Risk factor for aortic dissection in Chinese pupolation | Risk factor